CLINICAL TRIAL: NCT02989181
Title: Impact of Continues Positive Airway Pressure Treatment in Patients With Dilated Cardiomyopathy and Obstructive Sleep Apnea (RIDA)
Brief Title: Continues Positive Airway Pressure Treatment for Patients With Dilated Cardiomyopathy and Obstructive Sleep Apnea
Acronym: RIDA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Göteborg University (Other)
Responsible Party: Principal Investigator, Maria Schaufelberger, Associate Professor, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FoU127221
Record Dates: First submitted 2016-09-09; First posted 2016-12-12 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Dilated Cardiomyopathy; Obstructive Sleep Apnea
MeSH Terms: conditions — Cardiomyopathy, Dilated; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continues Positive Airway Pressure (Experimental): Use of Continues Positive Airway Pressure (CPAP) mask every night under six months period.
  Interventions: Device: Continues Positive Airway Pressure (CPAP)
- Consultation of conservative measures (No Intervention): Study participants with DCM and OSA (no-CPAP), participants receive consultation of conservative measures such as avoiding alcohol before bedrest, sleeping on the side...

INTERVENTIONS:
Device: Continues Positive Airway Pressure (CPAP) — Mask with positive airway pressure during exhalation which maintains the airway open
  Arms: Continues Positive Airway Pressure

SUMMARY:
The aim of this randomized controlled study is to investigate the effect of continues positive airway pressure (CPAP) treatment in patients with dilated cardiomyopathy (DCM) and concomitant obstructive sleep apnea (OSA). The primary endpoint is left ventricular function measured by magnetic resonance (improvement of at least 4%) after six months treatment with CPAP.

The secondary endpoints include diastolic dysfunction, cardiovascular biomarkers and quality of life.

DETAILED DESCRIPTION:
Sleep apnea, either obstructive (OSA) and central (CSA), occurs in more than half of all patients with heart failure (HF), and is associated with poor prognosis in these individuals.

Dilated cardiomyopathy (DCM) is the most common type of cardiomyopathy and is defined as the presence of the left ventricle dilatation and left ventricular systolic dysfunction without concurrent valvular or coronary artery disease. Its etiology is unclear, but a genetic component is present in at least 25% of cases. In younger individuals, the etiology is more heterogeneous, where a rare type of cardiomyopathy may occur in women in connection with pregnancy, s.c. peripartum cardiomyopathy. Other underlying causes include alcohol, drugs, pharmaceuticals, endocrine disorders, systemic diseases and general muscle. These factors account for approximately half the cases of DCM in younger and other half designated as idiopathic (IDCM).

The relationship between cardiomyopathies and OSA is insufficiently studied so far. In a smaller population of 20 individuals with DCM, sleep apnea (OSA or CSA) had 16, ie 80% of patients. The first-line treatment of OSA is continues positive pressure breathing mask (CPAP) during sleep in patients with daytime sleepiness. Effect of CPAP therapy in patients with DCM and OSA is completely unknown, because many of them do not report daytime sleepiness. The fact that patients with heart failure and reduced pumping function usually have symptoms of including fatigue, it becomes difficult to distinguish what is fatigue due to heart failure and what is related to sleep apnea. Interpretation of the Epworth Sleepiness Scale (ESS) is thus difficult and possibly unsure why all patients with DCM and OSA will be randomized to treatment with CPAP.

ELIGIBILITY:
Inclusion Criteria:

Patients with newly diagnosed or previously known DCM, treated and followed at cardiology outpatients clinic, stable in their symptoms and functional class at least 2 weeks after the last medicine change.

* Consent for the study.
* EF ≤ 45%.
* OSA diagnosis (Apnea-Hypopnea index> = 15 in the sleep recording below).

Exclusion Criteria:

* Patients already treated with Continues Positive Airway Pressure.
* Patients with claustrophobia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction (LVEF) six months after randomization to Continues Positive Airway Pressure (CPAP) treatment or consultation of conservative measures | 6 months
  The primary endpoint is left ventricular ejection fraction (LVEF) measured by cardiac magnetic resonance (improvement of at least 4%) at study baseline and at 6 months after randomization to Continues Positive Airway Pressure (CPAP) or consultation of conservative measures.
Change in left ventricular ejection fraction (LVEF) six months after randomization to Continues Positive Airway Pressure (CPAP) treatment or consultation of conservative measures | 6 months
  The primary endpoint is left ventricular ejection fraction (LVEF) measured by echocardiography at study baseline and at 6 months after randomization to Continues Positive Airway Pressure (CPAP) or consultation of conservative measures.

SECONDARY OUTCOMES:
Change in measurements of diastolic function after randomization to Continues Positive Airway Pressure (CPAP) or consultation of conservative measures. | baseline and at six months
  Secondary outcomes include measurements of diastolic function measured by cardiac magnetic resonance (CMR) and echocardiography,
Change in measurements of cardiovascular biomarkers at | baseline and at six months
  Analyzing change in cardiovascular biomarkers by analyzing blood samples
Change in quality of life questioners | baseline and at six months
  Analyzing participants response to quality of life by analyzing established questioners regarding dilated cardiomyopathy (Kansas city cardiomyopathy questionnaire KCCQ).
Change in day-time sleepiness | baseline and at six month
  Analyzing participants respons to established questioners regarding sleep apnea (Epworth sleepiness scale ESS) and

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital/Östra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided